CLINICAL TRIAL: NCT01023139
Title: "Efficacy in Adolescents of Continued Behavior Modification Following a Six Month Sibutramine-based Weight Management Intervention"
Acronym: AOS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Brooke Army Medical Center (U.S. Federal Agency)
Collaborators: 59th Medical Wing (U.S. Federal Agency)
Responsible Party: Jorge L. Cabrera, Brooke Army Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: c.2009.025
Record Dates: First submitted 2009-12-01; First posted 2009-12-02 (Estimated); Last update posted 2009-12-02 (Estimated); Status verified 2009-12

CONDITIONS: Obesity
Keywords: Adolescent; Obesity; Pharmacotherapy; Sibutramine
MeSH Terms: conditions — Obesity | interventions — sibutramine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard of care (SOC) (No Intervention): No intervention following phase 1 of the study is done during this 2nd phase. Participants will have their height and weights examined at 3 month and 6 month following end of phase 1. During these two visits, they will receive counseling from the physician regarding food choices and exercise maintenance.
- Continuing Behavioral Therapy (CoBT) (Experimental): This arm follows the end of the phase 1 which incorporates behavioral therapy, nutrition counseling and pharmacotherapy with Sibutramine while medically supervised. Participants randomized to this arm no longer receive medication and will receive behavioral therapy once a month and then evaluated at 3 months and six months for weight loss maintenance.
  Interventions: Behavioral: Sibutramine

INTERVENTIONS:
Behavioral: Sibutramine — During phase 1, sibutramine is given to all participants, 10mg po q day. If they do not meet a change in BMI of at least 2.5%,then the dosage may be increased to 15mg po q day. The main intervention in the study during phase 1 and 2is the behavioral modification
  Arms: Continuing Behavioral Therapy (CoBT)

SUMMARY:
There are few studies that look at sustained weight loss in the adolescent population. This study uses a multidisciplinary approach along with pharmacotherapy (use of Meridia)to motivate and establish behavior changes in adolescents (12-18yo) during the first phase of the study.

The second phase will have those who have lost at least 5% BMI to be randomized into one of two groups. This first group will have no intervention and will be followed at 3 and 6 months to assess for weight loss maintenance. The second group will continue on with monthly behavior modifications and also be evaluated at 3 and 6 months.

The hypothesis proposed is that, 1)there will be sustained weight loss at the end of one year in both arms as compared to baseline BMI, 2) and the arm with the behavioral therapy intervention will be more successful than no intervention at weight loss maintenance.

ELIGIBILITY:
Inclusion Criteria:

* Age: > or = 12 and < or = 18 years old at the time of screening

  * BMI that is at least more than the U.S. weighted mean of the 95th percentile based on age and sex
  * Willing to lose weight to meet and continue study medication for the 12 month treatment period even if he/she meets personal weight loss goal.
  * Willing to not start any new weight loss products
  * Males or non-pregnant females (pregnancy determined by self-report)
  * Females of childbearing potential if practicing acceptable method of contraception

Exclusion Criteria:

* Weight loss ≥ 10 pounds in previous 3 months
* Active gastrointestinal disorders (except GERD) such as peptic ulcer disease, irritable bowel disease, and gallbladder condition (in last 3 months); inflammable bowel disease (Crohn's ulcerative colitis, celiac sprue)
* At least 2 out of 3 blood pressure readings either systolic or diastolic ≥ 95%ile for height and age or pulse ≥95 beats per minute at initial visit.
* Drug treated diabetes mellitus or drug treated hypertension
* Drugs and/or supplements administered for the first time or withdrawn during the past 6 months which have a significant impact on body weight or digestion (see Appendix D)
* Inability or unwillingness to comply with protocol requirements, i.e. considered to be unfit for study participation, or unable to swallow pills.
* Unwilling to avoid consumption of alcoholic beverages
* Smoking or has started a smoking cessation program within the past six months
* Previous treatment with prescription sibutramine (Meridia®)
* History of recurrent nephrolithiasis
* Major psychiatric or eating disorders (i.e., major depressive disorder, bipolar disorder, anorexia nervosa, bulimia or laxative abuse)
* Kidney, liver, or thyroid disorder
* Drugs that are contraindicated with concomitant use of sibutramine (Meridia®) within last 4 weeks (See Appendix E)
* Cardiovascular disease (including arrhythmias, heart failure or congenital heart defect
* History of bleeding problems, hemophilia
* History of migraine headaches; seizures; a stroke or mini-stroke
* History of Pulmonary hypertension
* Osteopenia or osteoporosis
* Self-report of current recreational drug use or overused prescription medications
* History of glaucoma
* Females who self-report pregnancy

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2009-04; Primary Completion 2010-11 (Estimated); Study Completion 2011-03 (Estimated)

PRIMARY OUTCOMES:
% change in BMI z score | 12 month

SECONDARY OUTCOMES:
absolute weight change | 12 months
waist circumference change | 12 month

CONTACTS AND LOCATIONS:
Overall Officials: Jorge L Cabrera, MD, PhD, Principal Investigator — Brooke Army Medical Center
Locations (2):
- United States (2):
  - Brooke Army Medical Center, San Antonio, Texas
  - Wilford Hall Medical Center, San Antonio, Texas